CLINICAL TRIAL: NCT05395299
Title: Feasibility of Prostatic Arterial Embolization With SQUID (Ethylene Vinyl Alcohol Copolymer ) in Symptomatic Patients With Benign Prostatic Hyperplasia: Monocentric Pilot Study
Brief Title: Prostatic Arterial Embolization With SQUID (Ethylene Vinyl Alcohol Copolymer )
Acronym: SQUID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-PP-21; 2021-A02956-35 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-04-29; First posted 2022-05-27 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Prostatic Hyperplasia, Benign
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — ethylene-vinyl alcohol copolymer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prostatic Arterial Embolization with SQUID (Ethylene Vinyl Alcohol Copolymer ) (Experimental): Injection at the level of the right and left prostate arteries of Squid until a complete occlusion of these arteries, and a filling of their intraprostatic branches
  Interventions: Procedure: SQUID (Ethylene Vinyl Alcohol Copolymer ) administred to the participant with the intervention Prostatic Arterial Embolization

INTERVENTIONS:
Procedure: SQUID (Ethylene Vinyl Alcohol Copolymer ) administred to the participant with the intervention Prostatic Arterial Embolization — Prostatic Arterial Embolization with SQUID (Ethylene Vinyl Alcohol Copolymer )

SUMMARY:
The aim of this pilot study is to analyze the feasibility of prostatic embolization for the treatment of symptomatic benign prostatic hypertrophy with a non adhesive liquid embolic agent (Squid)

DETAILED DESCRIPTION:
Microparticle prostatic embolization is an effective technique in the short and medium term in the treatment of symptoms related to benign prostatic hyperplasia. If this technique allows an improvement of the patients' symptoms, and fewer operative complications than urological interventions, on the other hand, the injection of arterial particles has several disadvantages: a random long-term durability mainly due to a revascularization of the embolized territories ; inferiority compared to urological treatments in terms of reduction of prostate volume and improvement of postoperative urodynamic tests; poor visualization of the embolization material, and a risk of injection of the particles into an artery supplying a non-target organ. Ethylene vinyl alcohol copolymer is a liquid embolism used for the endovascular treatment of cerebral arteriovenous malformations since 2005 and in specific extracerebral applications due to its advantageous physical properties (its viscous nature, its slow polymerization, its definitive and very distal occlusion, and its high fluoroscopic visibility). These properties would allow in prostatic embolization: to obtain better control during the injection and therefore to improve the safety of the embolization; to reduce the risk of recurrence; and to achieve a more intense prostatic ischemia and therefore to obtain a greater reduction in prostatic volume, and a better improvement in urodynamic tests. The aim of this pilot study is to analyze the feasibility of injecting this liquid embolic agent during the endovascular treatment of symptomatic benign prostatic hypertrophy. If this preliminary study is positive, a randomized phase III study could be undertaken to judge the results and the place of this technique in the treatment of symptoms related to benign prostatic hyperplasia.

ELIGIBILITY:
Inclusion Criteria

* Patient over 45 and under 80
* Benign prostatic hypertrophy with an obstructive syndrome of the lower urinary tract intolerant or refractory to medical treatment (continued for 6 months)
* Indication of prostatic embolization.
* Prostate volume of more than 40 ml

  - Subject with an IPSS> 18 and a Qol> 3
* Affiliation to a social security scheme.
* Subject who has given informed consent to participate in the study.

Exclusion criteria patient with prostate cancer or suspected of having prostate cancer

* patient with neurological bladder or AUS of extra-prostatic origin
* detrusor dysfunction
* documented allergy to iodinated contrast media
* Hepatic insufficiency
* advanced arteritis
* severe renal failure with glomerular filtration rate <60 ml / min / 1.73 m2 body surface area
* inability to independently complete the self-questionnaires used in the study • acute or chronic prostatitis
* hydronephrosis
* diverticulum larger than 2 cm or bladder calculus
* ureteral stenosis
* active infectious syndrome
* major surgery in the four months preceding the inclusion visit
* Progressive cancer or for which the risk of progressive recovery is more than 50% in the next 5 years
* limited life expectancy
* Vulnerable persons defined in Articles L. 1121-5 to L.1121-8 and L.1122-1-2 of the Public Health Code (eg: persons deprived of their liberty, minors, protected adults, etc.)

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2024-10-05 (Actual)

PRIMARY OUTCOMES:
The main objective is to study the feasibility of prostate embolization with SQUID | day 0
  squid injection success in the prostate assessed by a scanner

SECONDARY OUTCOMES:
Description of the causes of technical embolization failures | day 0
  Injection into the 2 prostate lobes

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sedat J, Fontas E, Arnoffi P, Stranieri G, Colomb F, Chau Y. Prostatic Artery Embolization Using Ethylene Vinyl Alcohol (EVOH) Copolymer for Benign Prostatic Hyperplasia: Twelve-Month Analysis. Cardiovasc Intervent Radiol. 2025 Sep;48(9):1369-1375. doi: 10.1007/s00270-025-04164-x. Epub 2025 Aug 13. PMID 40804546
- [Derived] Sedat J, Arnoffi P, Poirier F, Jamjoom M, Raffaelli C, Colomb F, Chau Y. Non-target embolic events during prostatic embolization with ethylene vinyl alcohol copolymer (EVOH). CVIR Endovasc. 2023 Nov 3;6(1):54. doi: 10.1186/s42155-023-00402-w. PMID 37922055